CLINICAL TRIAL: NCT05552274
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Repeated Dose Escalation, FTIH Study to Investigate the Safety, Tolerability, PK and PD of ECC4703 in Healthy Volunteers and Participants With Treatment-Unnecessary LDL-C Under 160 mg/dL
Brief Title: FTIH of ECC4703 in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC0002
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAD Cohorts 1 to 2: Participants receiving Placebo (Placebo Comparator): Participants in each SAD cohort will be randomized to receive placebo
  Interventions: Drug: Placebo
- SAD Cohorts 1 to 2: Participants receiving ECC4703 (Experimental): Participants in each SAD cohort will be randomized to receive up to 4 escalating doses (1 mg, 4 mg, 12 mg, 32 mg, 80 mg, 160 mg, 320 mg or 400 mg).
  Interventions: Drug: ECC4703
- MAD Cohorts 1 to 4: Participants receiving Placebo (Placebo Comparator): Participants will be randomized to receive a once-daily dose of placebo for 14 days.
  Interventions: Drug: Placebo
- MAD Cohorts 1 to 4: Participants receiving ECC4703 (Experimental): Participants will be randomized to receive a once-daily dose of 1 of 3 escalating doses (40 mg, 80 mg, or 160 mg) for 14 days.
  Interventions: Drug: ECC4703

INTERVENTIONS:
Drug: ECC4703 — ECC4703 will be administered as 1 mg, 10 mg and 40 mg capsules. ECC4703 will be administered as oral capsules during each dosing day.
  Arms: MAD Cohorts 1 to 4: Participants receiving ECC4703; SAD Cohorts 1 to 2: Participants receiving ECC4703
Drug: Placebo — Matching Placebo will be administered as oral capsules. Matching Placebo will be given orally during each dosing day.
  Arms: MAD Cohorts 1 to 4: Participants receiving Placebo; SAD Cohorts 1 to 2: Participants receiving Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose and multiple ascending dose study of ECC4703 in healthy volunteers and participants with treatment unnecessary LDL-C under 160 mg/dL

DETAILED DESCRIPTION:
This study will be conducted in two cohorts of Single Ascending Dose (SAD) with a dose range from 1mg to 400mg and in four cohorts of Multiple Ascending Dose (MAD) with a dose range of 40mg to 160mg to Investigate the Safety, Tolerability, PK, and PD of ECC4703 in Healthy Volunteers and Participants with Treatment Unnecessary LDL-C under 160 mg/dL

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants of any ethnic origin
* Age of 18 to 65 years
* BMI of 18.0 to 32.0 kg/m2
* Female participants who are postmenopausal, confirmed by FSH test, or surgically sterile, confirmed by medical documentation, or if they are of child bearing potential agree to use at least 1 highly effective method of contraception and 1 additional effective method at the same time, or agree to practice true abstinence
* Male participants agree to use contraception, or agree to practice true abstinence
* No clinically significant findings in physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, laboratory tests, or medical/psychiatric history
* Not taking any medication on a regular basis
* Able to understand and sign and date informed consent

Additional Inclusion Criteria for Part 2 (MAD) Cohorts B2 to B4

* Fasting LDL-C ≥ 100 mg/dL and ≤ 159 mg/dL at screening
* Not eligible for lipid-lowering therapy (such as statin) as decided by the qualified clinician at screening based on <2019 ACC/AHA Guidelines on the Primary Prevention of Cardiovascular Disease>
* Hemoglobin A1c (HbA1c) ≤ 6.5%.

Exclusion Criteria:

* Females who are pregnant including a positive result of pregnancy test, planning to become pregnant, or breastfeeding.
* History of febrile illness or evidence of active infection within 14 days prior to the first dose of study;
* Use of any concomitant medication
* History of drug abuse or alcohol abuse within the past 5 years;
* Regular use of tobacco, nicotine or tobacco products within the past 6 months of the study ;
* Unwilling to abstain from alcohol containing products and/or xanthine/caffeine containing products, including any food and beverages, within 48 h prior to the first dose of study drug;
* Concomitant participation in any investigational study of any nature
* Blood loss of non-physiological reasons ≥ 200 ml (i.e. trauma, blood collection, blood donation) within 2 months prior to the first dose of study drug, or plan to donate blood during this trial and within 1 month after the last dosing;
* Abnormal renal function estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m2
* Currently diagnosed type 2 diabetes mellitus (T2DM) or has history of T2DM.
* Significant allergic reaction to active ingredients or excipients of the study drug.
* Any clinically significant abnormal findings in the participant's physical examination, laboratory tests, pregnancy test, urine drug screen, alcohol test, or medical history which in the opinion of the Investigator would prevent the participants from participating in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events, with abnormal laboratory test results, abnormal ECGs, abnormal vital signs, and abnormal physical examinations | SAD: Up to 8 days and MAD: Up to 21 days
  Safety Assessment evaluated through adverse events, laboratory evaluations, vital signs, ECGs, and physical examination.

SECONDARY OUTCOMES:
Pharmacokinetic Parameters: AUC0-24 | SAD: Up to Day 8 and MAD: Up to Day 21.
  AUC from time 0 to 24 hour dosing interval
Pharmacokinetic Parameters: AUC0-tlast | SAD: Up to Day 8
  AUC from time 0 to the time of last quantifiable non-zero concentration
Pharmacokinetic Parameters: AUC0-tau | MAD: Up to Day 21.
  AUC over a dosing interval from time 0 to time of last quantifiable concentration
Pharmacokinetic Parameters: AUC0-infinity | SAD: Up to Day 8
  AUC from time 0 extrapolated to infinity
Pharmacokinetic Parameters: Cmax | SAD: Up to Day 8 and MAD: Up to Day 21.
  Maximum observed plasma concentration
Pharmacokinetic Parameters: C24 | SAD: Up to Day 8 and MAD: Up to Day 21.
  Observed concentration at 24 hours post dose
Pharmacokinetic Parameters: Ctau | MAD: Up to Day 21.
  Observed concentration at the end of the dosing interval
Pharmacokinetic Parameters: tmax | SAD: Up to Day 8 and MAD: Up to Day 21.
  Time of the maximum observed plasma concentration
Pharmacokinetic Parameters: tlag | SAD: Up to Day 8 and MAD: Up to Day 21.
  Lag time (time delay between dosing and first observed plasma concentration)
Pharmacokinetic Parameters: t1/2 | SAD: Up to Day 8 and MAD: Up to Day 21.
  Apparent terminal elimination half-life
Pharmacokinetic Parameters: Clast | SAD: Up to Day 8
  Last measurable non-zero concentration
Pharmacokinetic Parameters: tlast | SAD: Up to Day 8
  Time of last measurable non-zero concentration
Pharmacokinetic Parameters: CL/F | SAD: Up to Day 8 and MAD: Up to Day 21.
  Apparent Clearance
Pharmacodynamic assessment: LDL-C | SAD: Up to Day 8
  Measurement of Low Density Lipoprotein Cholesterol
Pharmacodynamic assessment: HDL-C | MAD: Up to Day 21.
  Measurement of High Density Lipoprotein Cholesterol
Pharmacodynamic assessment: TG | MAD: Up to Day 21.
  Measurement of Triglycerides
Pharmacodynamic assessment: TC | MAD: Up to Day 21.
  Measurement of Total Cholesterol
Pharmacodynamic assessment: LDL | MAD: Up to Day 21.
  Measurement of Low Density Lipoprotein
Pharmacodynamic assessment: VLDL | MAD: Up to Day 21.
  Measurement of Very Low Density Lipoprotein
Pharmacodynamic assessment: ApoB | SAD: Up to Day 8 and MAD: Up to Day 21.
  Measurement of Apolipoprotein B
Pharmacodynamic assessment: Lp(a) | MAD: Up to Day 21.
  Measurement of Lipoprotein (a)
Pharmacodynamic assessment: Glucose | MAD: Up to Day 21.
  Measurement of Glucose
Pharmacodynamic assessment: Serum Insulin | MAD: Up to Day 21.
  Measurement of Serum Insulin
Thyroid function assessment: TT3 | SAD: Up to Day 8 and MAD: Up to Day 21.
  Measurement of Total Triiodothyronine
Thyroid function assessment: FT3 | SAD: Up to Day 8 and MAD: Up to Day 21.
  Measurement of Free Triiodothyronine
Thyroid function assessment: TT4 | SAD: Up to Day 8 and MAD: Up to Day 21.
  Measurement of Total Thyroxine
Thyroid function assessment: FT4 | SAD: Up to Day 8 and MAD: Up to Day 21.
  Measurement of Free Thyroxine
Thyroid function assessment: TSH | SAD: Up to Day 8 and MAD: Up to Day 21.
  Measurement of Thyroid Stimulating Hormone

CONTACTS AND LOCATIONS:
Overall Officials: Eccogene, Study Director — Eccogene Clinical Trials
Locations (1):
- Eccogene Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No